CLINICAL TRIAL: NCT01323946
Title: Safety and Immunogenicity of GSK Biologicals' (Pre-) Pandemic Influenza Candidate Vaccine (GSK1562902A) in Children Aged 6 to 35 Months
Brief Title: Study to Evaluate the Immunogenicity and Safety of an Investigational Pandemic Influenza Vaccine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109825; 2011-004734-33 (EudraCT Number)
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Influenza
Keywords: H5N1; influenza infection; Influenza vaccine GSK1562902A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Subjects were to be stratified into three age strata (6 to 11 months, 12 to 23 months and 24 to 35 months) in the ratio of 2:1:1.

ARMS (3):
- GSK1562902A 6 to 12 M Group (Experimental): Subjects between 6 and 12 months of age (6 to 12 M), who received 2 primary doses of A/Indonesia/05/2005 GSK1562902A vaccine on Days 0 and 21 and 1 booster dose of the A/turkey/Turkey/1/2005 GSK1562902A vaccine on Day 182.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK1562902A
- GSK1562902A 12 to 24 M Group (Experimental): Subjects between 12 and 24 months of age (12 to 24 M), who received 2 primary doses of A/Indonesia/05/2005 GSK1562902A vaccine on Days 0 and 21 and 1 booster dose of the A/turkey/Turkey/1/2005 GSK1562902A vaccine on Day 182.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK1562902A
- GSK1562902A 24 to 36 M Group (Experimental): Subjects between 24 and 36 months of age (24 to 36 M), who received 2 primary doses of A/Indonesia/05/2005 GSK1562902A vaccine on Days 0 and 21 and 1 booster dose of the A/turkey/Turkey/1/2005 GSK1562902A vaccine on Day 182.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK1562902A

INTERVENTIONS:
Biological: GSK Biologicals' investigational vaccine GSK1562902A — Three intramuscular injections

SUMMARY:
The objective of the study is to evaluate the immunogenicity and safety of prime-boost vaccination schedule of GSK Biologicals' investigational vaccine GSK1562902A.

DETAILED DESCRIPTION:
This protocol posting was modified according to the protocol amendment 2 (dated 16-June-2011). The impacted section is eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parents/Legally Acceptable Representatives (LARs) can and will comply with the requirements of the protocol.
* Children, male or female between, and including, 6 and 35 months of age at the time of first study vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy children as established by medical history and clinical examination before entering the study.
* Parent/LAR access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device.
* Subjects who are likely to reside in the vicinity of the study centre for the duration of the study. In studies using the home-based model for vaccination and follow-up, subjects who are likely to remain in the vicinity of the area where they were recruited.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration of any vaccine 30 days prior and 21 days after any study vaccine administration.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines such as egg protein or thiomersal.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any neurological disorders or seizures.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory tests.
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study, or planned administration during the study period.
* Any condition which, in the opinion of the investigator, renders the subject unfit for participation in the study.
* Child in care.
* Previous vaccination at any time with an H5N1 vaccine.
* Medical history of physician-confirmed infection with a H5N1 virus.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2011-04-18 (Actual); Primary Completion 2012-06-22 (Actual); Study Completion 2012-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Australia (4):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Carlton, Victoria
- GSK Investigational Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Nolan T, Izurieta P, Lee BW, Chan PC, Marshall H, Booy R, Drame M, Vaughn DW. Heterologous prime-boost vaccination using an AS03B-adjuvanted influenza A(H5N1) vaccine in infants and children<3 years of age. J Infect Dis. 2014 Dec 1;210(11):1800-10. doi: 10.1093/infdis/jiu359. Epub 2014 Jun 27. PMID 24973461
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 109825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109825 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/ exclusion criteria, contraindications/ precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group
Started | 46 | 34 | 33
Completed | 43 | 31 | 33
Not Completed | 3 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Parents refused the last blood draw | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | Total
Number analyzed (Participants) | 46 | 34 | 33 | 113
Age, Continuous [Mean (Standard Deviation); unit: Months] | 8.3 (1.56) | 16.1 (3.44) | 29.6 (3.38) | 16.87 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 19 | 63
  Male | 21 | 15 | 14 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian -South East Asian heritage, n(%) | 33 | 25 | 22 | 80
  Asian - east asian heritage | 0 | 1 | 0 | 1
  White - caucasian / european heritage | 12 | 8 | 9 | 29
  Unspecified | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects in Terms of H5N1 Hemagglutination Inhibition (HI) Antibodies Against A/Turkey/Turkey/1/2005 H5N1 Virus Strain
Description: A seroconverted subject is defined as a subject that had either a pre-vaccination (Day 0) titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer on Day 192.
Time Frame: At Day 192
Population: The analysis was performed on the ATP cohort for immunogenicity at Month 6, including all evaluable subjects for whom considered assay results were available for pre-vaccination (Day 0) and post-vaccination (Day 192) time points. Analyses were done by age stratum and overall.
Measure: Count of Participants; unit: Participants
Groups:
- GSK1562902A Group: Subjects received 2 primary doses of A/Indonesia/05/2005 GSK1562902A vaccine on Days 0 and 21 and 1 booster dose of the A/turkey/Turkey/1/2005 GSK1562902A vaccine on Day 182.
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 33 | 21 | 29 | 83
Participants | 33 | 21 | 29 | 83

2. Primary Outcome: Mean Geometric Change in Terms of H5N1 HI Antibodies Against A/Turkey/Turkey/01/2005 H5N1 Virus Strain
Description: Mean Geometric Change is defined as the geometric mean of the within-subject ratios of the post vaccination (Day 192) reciprocal HI titer to the pre-vaccination (Day 0) reciprocal HI titer (i.e. post-vaccination divided by pre-vaccination titer).
Time Frame: At Day 192
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- GSK1562902A Group: Subjects received 2 primary doses of A/Indonesia/05/2005 GSK1562902A vaccine on Days 0 and 21 and 1 booster dose of the A/turkey/Turkey/1/2005 H5N1 vaccine on Day 182.
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 33 | 21 | 29 | 83
Titers | 424.1 [327.3 to 549.4] | 317.6 [208.4 to 484.0] | 321.2 [248.4 to 415.5] | 357.7 [302.4 to 423.2]

3. Primary Outcome: Number of Seroprotected Subjects in Terms of H5N1 HI Antibodies Against A/Turkey/Turkey/01/2005 H5N1 Virus Strain
Description: A seroprotected subject is defined as a subject with a serum H5N1 HI antibody titer ≥1:40.
Time Frame: At Day 192
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 33 | 21 | 29 | 83
Participants | 33 | 21 | 29 | 83

4. Secondary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against the A/Indonesia/05/2005 H5N1 Virus Strain
Description: Titers were presented as geometric mean titers (GMTs). Analyses were done by age stratum and overall.
Time Frame: At Day 0, Day 42, Day 182, Day 192 and Day 364
Population: The analysis was performed on the ATP cohort for immunogenicity at Month 6 (Day 0, 42, 182 and 192) and Month 12 (Day 364), including all evaluable subjects for whom considered assay results were available for the considered time point. Analyses were done by age stratum and overall.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 27 | 32 | 100
Titer
  A/Indonesia/05/2005.HA [Day 0]: number analyzed (Participants) | 33 | 24 | 29 | 86
  A/Indonesia/05/2005.HA [Day 0] | NA [NA to NA] — GMTs could not be computed as none of the subjects had HI antibody titers above the assay cut-off value of 1:10. | NA [NA to NA] — GMTs could not be computed as none of the subjects had HI antibody titers above the assay cut-off value of 1:10. | NA [NA to NA] — GMTs could not be computed as none of the subjects had HI antibody titers above the assay cut-off value of 1:10. | NA [NA to NA] — GMTs could not be computed as none of the subjects had HI antibody titers above the assay cut-off value of 1:10.
  A/Indonesia/05/2005.HA [Day 42]: number analyzed (Participants) | 32 | 24 | 29 | 85
  A/Indonesia/05/2005.HA [Day 42] | 945.2 [745.8 to 1197.9] | 1336.7 [990.3 to 1804.2] | 1044.7 [832.6 to 1310.9] | 1078.6 [935.3 to 1243.7]
  A/Indonesia/05/2005.HA [Day 182]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/Indonesia/05/2005.HA [Day 182] | 160.0 [125.4 to 204.2] | 147.3 [113.2 to 191.7] | 133.7 [113.1 to 158.1] | 147.2 [129.6 to 167.1]
  A/Indonesia/05/2005.HA [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/Indonesia/05/2005.HA [Day 192] | 2163.9 [1772.7 to 2641.4] | 1534.7 [1108.1 to 2125.5] | 1606.2 [1254.3 to 2056.9] | 1787.6 [1552.4 to 2058.3]
  A/Indonesia/05/2005.HA [Day 364] | 1465.4 [1168.2 to 1838.1] | 1055.8 [769.2 to 1449.1] | 668.4 [505.2 to 884.2] | 1043.3 [886.1 to 1228.4]

5. Secondary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against the A/Turkey/Turkey/01/2005 H5N1 Virus Strain
Description: Titers were presented as geometric mean titers (GMTs). Analyses were done by age stratum and overall.
Time Frame: At Day 0, Day 182, Day 192 and Day 364
Population: The analysis was performed on the ATP cohort for immunogenicity at Month 6 (Day 0, 182 and 192) and Month 12 (Day 364), including all evaluable subjects for whom considered assay results were available for the considered time point. Analyses were done by age stratum and overall.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 27 | 32 | 100
Titer
  A/turkey/Turkey/01/2005.HA [Day 0]: number analyzed (Participants) | 33 | 24 | 29 | 86
  A/turkey/Turkey/01/2005.HA [Day 0] | 5.8 [5.2 to 6.5] | 5.8 [4.8 to 6.9] | 5.5 [4.7 to 6.4] | 5.7 [5.2 to 6.2]
  A/turkey/Turkey/01/2005.HA [Day 182]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/turkey/Turkey/01/2005.HA [Day 182] | 95.7 [75.5 to 121.1] | 84.1 [65.5 to 108.1] | 86.1 [73.8 to 100.4] | 89.3 [79.1 to 100.7]
  A/turkey/Turkey/01/2005.HA [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/turkey/Turkey/01/2005.HA [Day 192] | 2454.6 [1935.7 to 3112.6] | 1810.2 [1207.1 to 2714.7] | 1767.4 [1403.0 to 2226.3] | 2026.2 [1731.3 to 2371.3]
  A/turkey/Turkey/01/2005.HA [Day 364] | 1810.1 [1466.6 to 2234.0] | 1263.8 [929.1 to 1719.0] | 803.4 [609.7 to 1058.8] | 1266.8 [1080.6 to 1485.0]

6. Secondary Outcome: Number of Seropositive Subjects in Terms of H5N1 HI Antibodies Against A/Indonesia/05/2005
Description: A seropositive subject is defined as a subject with a serum H5N1 HI antibody titer ≥ 1:10.
Time Frame: At Day 0, Day 42, Day 182, Day 192 and Day 364
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 27 | 32 | 100
Participants
  A/Indonesia/05/2005.HA [Day 0]: number analyzed (Participants) | 33 | 24 | 29 | 86
  A/Indonesia/05/2005.HA [Day 0] | 0 | 0 | 0 | 0
  A/Indonesia/05/2005.HA [Day 42]: number analyzed (Participants) | 32 | 24 | 29 | 85
  A/Indonesia/05/2005.HA [Day 42] | 32 | 24 | 29 | 85
  A/Indonesia/05/2005.HA [Day 182]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/Indonesia/05/2005.HA [Day 182] | 33 | 21 | 29 | 83
  A/Indonesia/05/2005.HA [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/Indonesia/05/2005.HA [Day 192] | 33 | 21 | 29 | 83
  A/Indonesia/05/2005.HA [Day 364] | 41 | 27 | 32 | 100

7. Secondary Outcome: Number of Seropositive Subjects in Terms of H5N1 HI Antibodies Against A/Turkey/Turkey/1/2005 H5N1 Virus Strain
Description: A seropositive subject is defined as a subject with a serum H5N1 HI antibody titer ≥ 1:10.
Time Frame: At Day 0, Day 182, Day 192 and Day 364
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 27 | 32 | 100
Participants
  A/turkey/Turkey/01/2005.HA [Day 0]: number analyzed (Participants) | 33 | 24 | 29 | 86
  A/turkey/Turkey/01/2005.HA [Day 0] | 6 | 3 | 2 | 11
  A/turkey/Turkey/01/2005.HA [Day 182] 83: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/turkey/Turkey/01/2005.HA [Day 182] 83 | 33 | 21 | 29 | 83
  A/turkey/Turkey/01/2005.HA [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/turkey/Turkey/01/2005.HA [Day 192] | 33 | 21 | 29 | 83
  A/turkey/Turkey/01/2005.HA [Day 364] | 41 | 27 | 32 | 100

8. Secondary Outcome: Number of Seroconverted Subjects in Terms of H5N1 HI Antibodies Against A/Indonesia/05/2005 H5N1 Virus Strain
Description: A seroconverted subjects is defined as a subject who had either a pre vaccination (Day 0) titer <1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Day 42, Day 182, Day 192 and Day 364
Population: The analysis was performed on the ATP cohort for immunogenicity at Month 6 (Day 42, 182 and 192) and Month 12 (Day 364), including all evaluable subjects for whom considered assay results were available for the pre-vaccination time point (Day 0) and the considered time point. Analyses were done by age stratum and overall.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 27 | 32 | 100
Participants
  A/Indonesia/05/2005.HA [Day 42]: number analyzed (Participants) | 32 | 24 | 29 | 85
  A/Indonesia/05/2005.HA [Day 42] | 32 | 24 | 29 | 85
  A/Indonesia/05/2005.HA [Day 182]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/Indonesia/05/2005.HA [Day 182] | 32 | 21 | 29 | 82
  A/Indonesia/05/2005.HA [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/Indonesia/05/2005.HA [Day 192] | 33 | 21 | 29 | 83
  A/Indonesia/05/2005.HA [Day 364] | 41 | 27 | 32 | 100

9. Secondary Outcome: Number of Seroconverted Subjects in Terms of H5N1 HI Antibodies Against A/Turkey/Turkey/1/2005 H5N1 Virus Strain
Description: A seroconverted subjects is defined as a subject who had either a pre vaccination (Day 0) titer <1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a 4-fold increase in post-vaccination titer. Data for Day 192 are presented under Primary Outcome Measures.
Time Frame: At Day 182 and Day 364
Population: The analysis was performed on the ATP cohort for immunogenicity at Month 6 (Day 182) and Month 12 (Day 364), including all evaluable subjects for whom considered assay results were available for the pre-vaccination time point (Day 0) and the considered time point. Analyses were done by age stratum and overall.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 26 | 32 | 99
Participants
  A/turkey/Turkey/1/2005 H5N1 (Day 182): number analyzed (Participants) | 33 | 21 | 29 | 83
  A/turkey/Turkey/1/2005 H5N1 (Day 182) | 31 | 20 | 28 | 83
  A/turkey/Turkey/1/2005 H5N1 (Day 364) | 41 | 26 | 28 | 95

10. Secondary Outcome: Number of Seroprotected Subjects in Terms of H5N1 HI Antibodies Against A/Indonesia/05/2005 Virus Strain
Description: A seroprotected subject is defined as a subject with a serum H5N1 HI antibody titer ≥1:40.
Time Frame: At Day 0, Day 42, Day 182, Day 192 and Day 364
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 27 | 32 | 100
Participants
  A/Indonesia/05/2005 H5N1.HA [Day 0]: number analyzed (Participants) | 33 | 24 | 29 | 86
  A/Indonesia/05/2005 H5N1.HA [Day 0] | 0 | 0 | 0 | 0
  A/Indonesia/05/2005 H5N1.HA [Day 42]: number analyzed (Participants) | 32 | 24 | 29 | 85
  A/Indonesia/05/2005 H5N1.HA [Day 42] | 32 | 24 | 29 | 85
  A/Indonesia/05/2005 H5N1.HA [Day 182]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/Indonesia/05/2005 H5N1.HA [Day 182] | 32 | 21 | 29 | 82
  A/Indonesia/05/2005 H5N1.HA [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/Indonesia/05/2005 H5N1.HA [Day 192] | 33 | 21 | 29 | 83
  A/Indonesia/05/2005 H5N1.HA [Day 364] | 41 | 27 | 32 | 100

11. Secondary Outcome: Number of Seroprotected Subjects in Terms of H5N1 HI Antibodies Against A/Turkey/Turkey/1/2005 H5N1 Virus Strain
Description: A seroprotected subject is defined as a subject with a serum H5N1 HI antibody titer ≥1:40. Data for Day 192 are presented under Primary Outcome Measures.
Time Frame: Day 0, Day 182 and Day 364
Population: The analysis was performed on the ATP cohort for immunogenicity at Month 6 (Day 0 and Day 182) and Month 12 (Day 364), including all evaluable subjects for whom considered assay results were available for the considered time point. Analyses were done by age stratum and overall.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 27 | 32 | 100
Participants
  A/turkey/Turkey/1/2005 H5N1.HA [Day 0]: number analyzed (Participants) | 33 | 24 | 29 | 86
  A/turkey/Turkey/1/2005 H5N1.HA [Day 0] | 0 | 0 | 1 | 1
  A/turkey/Turkey/1/2005 H5N1.HA [Day 182]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/turkey/Turkey/1/2005 H5N1.HA [Day 182] | 31 | 21 | 29 | 81
  A/turkey/Turkey/1/2005 H5N1.HA [Day 364] | 41 | 27 | 32 | 100

12. Secondary Outcome: Mean Geometric Change in Terms of H5N1 HI Antibodies Against A/Indonesia/05/2005 H5N1 Virus Strain
Description: Mean Geometric Change is defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination (Day 0) reciprocal HI titer (i.e. post-vaccination divided by pre-vaccination titer).
Time Frame: At Day 42, Day 182, Day 192 and Day 364
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 27 | 32 | 100
Titer
  A/Indonesia/05/2005 H5N1.HA [Day 42]: number analyzed (Participants) | 32 | 24 | 29 | 85
  A/Indonesia/05/2005 H5N1.HA [Day 42] | 189.0 [149.2 to 239.6] | 267.3 [198.1 to 360.8] | 208.9 [166.5 to 262.2] | 215.7 [187.1 to 248.7]
  A/Indonesia/05/2005 H5N1.HA [Day 182]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/Indonesia/05/2005 H5N1.HA [Day 182] | 32.0 [25.1 to 40.8] | 29.5 [22.6 to 38.3] | 26.7 [22.6 to 31.6] | 29.4 [25.9 to 33.4]
  A/Indonesia/05/2005 H5N1.HA [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/Indonesia/05/2005 H5N1.HA [Day 192] | 432.8 [354.5 to 528.3] | 306.9 [221.6 to 425.1] | 321.2 [250.9 to 411.4] | 357.5 [310.5 to 411.7]
  A/Indonesia/05/2005 H5N1.HA [Day 364] | 293.1 [233.6 to 367.6] | 211.2 [153.8 to 289.8] | 133.7 [101.0 to 176.8] | 208.7 [177.2 to 245.7]

13. Secondary Outcome: Mean Geometric Change in Terms of H5N1 HI Antibodies Against A/Turkey/Turkey/01/2005 H5N1 Virus Strain
Description: Mean Geometric Change is defined as the geometric mean of the within-subject ratios of the post vaccination reciprocal HI titer to the pre-vaccination (Day 0) reciprocal HI titer (i.e. post-vaccination divided by pre-vaccination titer). Data for Day 192 are presented under Primary Outcome Measures.
Time Frame: Day 182 and Day 364
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 26 | 32 | 99
Titer
  A/turkey/Turkey/1/2005 H5N1.HA [Day 182]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/turkey/Turkey/1/2005 H5N1.HA [Day 182] | 16.5 [12.8 to 21.4] | 14.8 [10.8 to 20.1] | 15.6 [12.5 to 19.5] | 15.8 [13.6 to 18.2]
  A/turkey/Turkey/1/2005 H5N1.HA [Day 364] | 19.9 [15.2 to 26.1] | 16.4 [12.6 to 21.4] | 9.5 [7.2 to 12.5] | 14.9 [12.6 to 17.6]

14. Secondary Outcome: Number of Booster Seroconverted Subjects in Terms of H5N1 HI Antibodies Against A/Turkey/Turkey/1/2005 H5N1 Virus Strain
Description: Booster seroconversion is defined as follows: For seronegative subjects at pre-booster (Day 182), antibody titer ≥1:40 at post-booster time point(s). For seropositive subjects at pre-booster (Day 182), antibody titer at post-booster time point(s) ≥4-fold the pre-booster antibody titer.
Time Frame: At Day 192 and Day 364
Population: The analysis was performed on the ATP cohort for immunogenicity at Month 6 (Day 192) and Month 12 (Day 364), including all evaluable subjects for whom considered assay results were available for the pre-booster vaccination time point (Day 182) and the considered time point. Analyses were done by age stratum and overall.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 26 | 32 | 99
Participants
  A/turkey/Turkey/01/2005 H5N1.HA [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/turkey/Turkey/01/2005 H5N1.HA [Day 192] | 32 | 21 | 29 | 82
  A/turkey/Turkey/01/2005 H5N1.HA [Day 364] | 41 | 26 | 28 | 95

15. Secondary Outcome: Booster Factor in Terms of Neutralizing Antibodies Against A/Turkey/Turkey/1/2005 H5N1 Virus Strain
Description: Booster Factor was defined as the geometric mean of the within-subject ratios of the post-booster vaccination reciprocal HI titer to the pre-booster (Day 182) reciprocal titer.
Time Frame: At Day 192 and Day 364
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 41 | 26 | 32 | 99
Titer
  A/turkey/Turkey/01/2005 H5N1.HA [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  A/turkey/Turkey/01/2005 H5N1.HA [Day 192] | 25.7 [18.4 to 35.7] | 21.5 [16.4 to 28.2] | 20.5 [16.2 to 26.1] | 22.7 [19.3 to 26.8]
  A/turkey/Turkey/01/2005 H5N1.HA [Day 364] | 19.9 [15.2 to 26.1] | 16.4 [12.6 to 21.4] | 9.5 [7.2 to 12.5] | 14.9 [12.6 to 17.6]

16. Secondary Outcome: Number of Seropositive Subjects in Terms of Serum Neutralizing Antibodies Against A/Indonesia/05/2005 H5N1 Virus Strain
Description: A seropositive subject is defined as a subject with serum neutralizing antibody titers ≥ 1:28
Time Frame: Day 0, Day 42, Day 182, Day 192 and Day 364
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 37 | 27 | 31 | 95
Participants
  Flu A/Ind/05/05 (H5N1) [Day 0]: number analyzed (Participants) | 29 | 22 | 24 | 75
  Flu A/Ind/05/05 (H5N1) [Day 0] | 0 | 0 | 1 | 1
  Flu A/Ind/05/05 (H5N1) [Day 42]: number analyzed (Participants) | 24 | 21 | 25 | 70
  Flu A/Ind/05/05 (H5N1) [Day 42] | 24 | 21 | 25 | 70
  Flu A/Ind/05/05 (H5N1) [Day 182]: number analyzed (Participants) | 32 | 21 | 28 | 81
  Flu A/Ind/05/05 (H5N1) [Day 182] | 32 | 21 | 28 | 81
  Flu A/Ind/05/05 (H5N1) [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  Flu A/Ind/05/05 (H5N1) [Day 192] | 33 | 21 | 29 | 83
  Flu A/Ind/05/05 (H5N1) [Day 364] | 37 | 27 | 31 | 95

17. Secondary Outcome: Number of Seropositive Subjects in Terms of Serum Neutralizing Antibodies Against A/Turkey/Turkey/1/2005 H5N1 Virus Strain
Description: A seropositive subject is defined as a subject with serum neutralizing antibody titers ≥ 1:28.
Time Frame: Day 0, Day 182, Day 192 and Day 364
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 37 | 27 | 31 | 95
Participants
  Flu A/Turk/01/05 (H5N1) [Day 0]: number analyzed (Participants) | 29 | 22 | 24 | 75
  Flu A/Turk/01/05 (H5N1) [Day 0] | 0 | 0 | 0 | 0
  Flu A/Turk/01/05 (H5N1) [Day 182]: number analyzed (Participants) | 32 | 21 | 28 | 81
  Flu A/Turk/01/05 (H5N1) [Day 182] | 32 | 21 | 28 | 81
  Flu A/Turk/01/05 (H5N1) [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  Flu A/Turk/01/05 (H5N1) [Day 192] | 33 | 21 | 29 | 83
  Flu A/Turk/01/05 (H5N1) [Day 364] | 37 | 27 | 31 | 95

18. Secondary Outcome: Serum Neutralizing Antibody Titers in Terms of Neutralizing Antibodies Against A/Indonesia/05/2005 H5N1 Virus Strain
Description: Titers were presented as geometric mean titers (GMTs).
Time Frame: Day 0, Day 42, Day 182, Day 192 and Day 364
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 37 | 27 | 31 | 95
Titer
  Flu A/Ind/05/05 (H5N1) [Day 0]: number analyzed (Participants) | 29 | 22 | 24 | 75
  Flu A/Ind/05/05 (H5N1) [Day 0] | NA [NA to NA] — Data could not be computed as none of the subjects had serum neutralizing antibody titers above the assay cut-off value of 1:28. | NA [NA to NA] — Data could not be computed as none of the subjects had serum neutralizing antibody titers above the assay cut-off value of 1:28. | 14.4 [13.6 to 15.3] | 14.1 [13.9 to 14.4]
  Flu A/Ind/05/05 (H5N1) [Day 42]: number analyzed (Participants) | 24 | 21 | 25 | 70
  Flu A/Ind/05/05 (H5N1) [Day 42] | 1785.9 [1168.6 to 2729.5] | 2080.4 [1422.8 to 3041.7] | 1755.2 [1191.3 to 2586.1] | 1858.0 [1491.3 to 2315.0]
  Flu A/Ind/05/05 (H5N1) [Day 182]: number analyzed (Participants) | 32 | 21 | 28 | 81
  Flu A/Ind/05/05 (H5N1) [Day 182] | 526.6 [397.1 to 698.2] | 483.3 [333.1 to 701.3] | 353.4 [273.7 to 456.2] | 448.7 [379.0 to 531.2]
  Flu A/Ind/05/05 (H5N1) [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  Flu A/Ind/05/05 (H5N1) [Day 192] | 12667.0 [10522.9 to 15248.1] | 11031.5 [8157.8 to 14917.5] | 9883.1 [7631.9 to 12798.4] | 11215.7 [9797.4 to 12839.2]
  Flu A/Ind/05/05 (H5N1) [Day 364] | 6420.9 [4851.0 to 8498.9] | 4730.9 [3237.5 to 6913.0] | 2422.9 [1674.9 to 3504.9] | 4283.3 [3485.8 to 5263.2]

19. Secondary Outcome: Serum Neutralizing Antibody Titers in Terms of Neutralizing Antibodies Against A/Turkey/Turkey/1/2005 H5N1 Virus Strain
Description: Titers were presented as geometric mean titers (GMTs).
Time Frame: Day 0, Day 182, Day 192 and Day 364
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 37 | 27 | 31 | 95
Titer
  Flu A/Turk/01/05 (H5N1) [Day 0]: number analyzed (Participants) | 29 | 22 | 24 | 75
  Flu A/Turk/01/05 (H5N1) [Day 0] | NA [NA to NA] — Data could not be computed as none of the subjects had serum neutralizing antibody titers above the assay cut-off value of 1:28. | NA [NA to NA] — Data could not be computed as none of the subjects had serum neutralizing antibody titers above the assay cut-off value of 1:28. | NA [NA to NA] — Data could not be computed as none of the subjects had serum neutralizing antibody titers above the assay cut-off value of 1:28. | NA [NA to NA] — Data could not be computed as none of the subjects had serum neutralizing antibody titers above the assay cut-off value of 1:28.
  Flu A/Turk/01/05 (H5N1) [Day 182]: number analyzed (Participants) | 32 | 21 | 28 | 81
  Flu A/Turk/01/05 (H5N1) [Day 182] | 137.5 [108.3 to 174.7] | 124.9 [104.3 to 149.5] | 113.2 [96.2 to 133.2] | 125.4 [111.6 to 140.8]
  Flu A/Turk/01/05 (H5N1) [Day 192]: number analyzed (Participants) | 33 | 21 | 29 | 83
  Flu A/Turk/01/05 (H5N1) [Day 192] | 7391.0 [5117.8 to 10674.0] | 5464.2 [3426.9 to 8712.7] | 3349.4 [2249.8 to 4986.4] | 5192.9 [4101.3 to 6575.1]
  Flu A/Turk/01/05 (H5N1) [Day 364] | 4149.7 [3028.8 to 5685.4] | 3030.8 [2036.2 to 4511.4] | 1317.8 [898.4 to 1933.0] | 2610.2 [2085.3 to 3267.2]

20. Secondary Outcome: Number of Subjects With a Vaccine Response in Terms of Serum Neutralizing Antibodies Against A/Indonesia/05/2005 H5N1 Virus Strain
Description: Vaccine response is defined as: For initially seronegative subjects, neutralizing antibody titer ≥ 1:56 at the considered time point after vaccination For initially seropositive subjects, neutralizing antibody titer ≥ 4 fold from pre-vaccination (Day 0)
Time Frame: At Day 42, Day 182, Day 192 and Day 364
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 33 | 25 | 25 | 83
Participants
  Flu A/Ind/05/05 (H5N1) [Day 42]: number analyzed (Participants) | 22 | 19 | 21 | 62
  Flu A/Ind/05/05 (H5N1) [Day 42] | 22 | 19 | 21 | 62
  Flu A/Ind/05/05 (H5N1) [Day 182]: number analyzed (Participants) | 28 | 19 | 23 | 70
  Flu A/Ind/05/05 (H5N1) [Day 182] | 28 | 19 | 22 | 69
  Flu A/Ind/05/05 (H5N1) [Day 192]: number analyzed (Participants) | 29 | 19 | 24 | 72
  Flu A/Ind/05/05 (H5N1) [Day 192] | 29 | 19 | 24 | 72
  Flu A/Ind/05/05 (H5N1) [Day 364] | 33 | 25 | 25 | 83

21. Secondary Outcome: Number of Subjects With a Vaccine Response in Terms of Serum Neutralizing Antibodies Against A/Turkey/Turkey/1/2005 H5N1 Virus Strain
Description: as for outcome 20
Time Frame: At Day 182, Day 192 and Day 364
Population: The analysis was performed on the ATP cohort for immunogenicity at Month 6 (Day 182 and 192) and Month 12 (Day 364), including all evaluable subjects for whom considered assay results were available for the pre-vaccination time point (Day 0) and the considered time point. Analyses were done by age stratum and overall.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 33 | 25 | 25 | 83
Participants
  Flu A/Turk/01/05 (H5N1) [Day 182]: number analyzed (Participants) | 28 | 19 | 23 | 70
  Flu A/Turk/01/05 (H5N1) [Day 182] | 22 | 17 | 19 | 58
  Flu A/Turk/01/05 (H5N1) [Day 192]: number analyzed (Participants) | 29 | 19 | 24 | 72
  Flu A/Turk/01/05 (H5N1) [Day 192] | 29 | 19 | 24 | 72
  Flu A/Turk/01/05 (H5N1) [Day 364] | 33 | 25 | 25 | 83

22. Secondary Outcome: Number of Subjects With a Booster Vaccine Response in Terms of Serum Neutralizing Antibodies Against A/Turkey/Turkey/1/2005 H5N1 Virus Strain
Description: Booster vaccine response is defined as: For seronegative subjects at Day 182, neutralizing antibody titers ≥ 1:56 at the considered time point after vaccination For seropositive subjects at Day 182, neutralizing antibody titers ≥ 4 fold from pre-vaccination (Day 182)
Time Frame: At Day 192 and Day 364
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 32 | 24 | 23 | 79
Participants
  Flu A/Turk/01/05 (H5N1) [Day 192]: number analyzed (Participants) | 28 | 19 | 23 | 70
  Flu A/Turk/01/05 (H5N1) [Day 192] | 27 | 19 | 23 | 69
  Flu A/Turk/01/05 (H5N1) [Day 364] | 32 | 22 | 22 | 76

23. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assigned were pain, swelling and redness. Any was defined as occurrence of any local symptom regardless of intensity grade; Grade 3 pain was defined as cried when limb was moved spontaneously painful.
Time Frame: During the 7-day post-vaccination period following each dose and across doses (Day 0 - Day 7, Day 21 - Day 28, Day 182 - Day 189)
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all subjects with at least one vaccine administration documented and with the symptom sheet filled-in. Analyses were done by age stratum and overall.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 46 | 33 | 33 | 112
Participants
  Any Pain Dose 1 | 14 | 5 | 13 | 32
  Grade 3 Pain Dose 1 | 2 | 0 | 1 | 3
  Any Redness Dose 1 | 2 | 0 | 2 | 4
  Grade 3 Redness Dose 1 | 0 | 0 | 0 | 0
  Any Swelling Dose 1 | 1 | 1 | 1 | 3
  Grade 3 Swelling Dose 1 | 0 | 0 | 0 | 0
  Any Pain Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Any Pain Dose 2 | 10 | 13 | 14 | 37
  Grade 3 Pain Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Grade 3 Pain Dose 2 | 0 | 0 | 1 | 1
  Any Redness Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Any Redness Dose 2 | 3 | 2 | 1 | 6
  Grade 3 Redness Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Grade 3 Redness Dose 2 | 0 | 0 | 0 | 0
  Any Swelling Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Any Swelling Dose 2 | 2 | 2 | 0 | 4
  Grade 3 Swelling Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Grade 3 Swelling Dose 2 | 0 | 0 | 0 | 0
  Any Pain Dose 3: number analyzed (Participants) | 45 | 33 | 33 | 108
  Any Pain Dose 3 | 20 | 15 | 18 | 53
  Grade 3 Pain Dose 3: number analyzed (Participants) | 45 | 33 | 33 | 108
  Grade 3 Pain Dose 3 | 3 | 1 | 3 | 7
  Any Redness Dose 3: number analyzed (Participants) | 45 | 33 | 33 | 108
  Any Redness Dose 3 | 11 | 5 | 2 | 18
  Grade 3 Redness Dose 3: number analyzed (Participants) | 45 | 33 | 33 | 108
  Grade 3 Redness Dose 3 | 0 | 0 | 0 | 0
  Any Swelling Dose 3: number analyzed (Participants) | 45 | 33 | 33 | 108
  Any Swelling Dose 3 | 5 | 5 | 1 | 11
  Grade 3 Swelling Dose 3: number analyzed (Participants) | 45 | 33 | 33 | 108
  Grade 3 Swelling Dose 3 | 0 | 0 | 0 | 0
  Any Pain Across doses | 26 | 19 | 21 | 66
  Grade 3 Pain Across doses | 4 | 1 | 5 | 10
  Any Redness Across doses | 13 | 6 | 3 | 22
  Grade 3 Redness Across doses | 0 | 0 | 0 | 0
  Any Swelling Across doses | 6 | 6 | 1 | 13
  Grade 3 Swelling Across doses | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were diarrhoea/ vomiting, drowsiness, irritability/ fussiness, loss of appetite, fever (axillary). Any= occurrence of any general symptom regardless of intensity grade and relationship to the vaccine. Irritability/ fussiness grade 3=crying that could not be comforted/ prevented normal activity; Drowsiness grade 3= drowsiness that prevented normal activity; Loss of appetite grade 3= did not eat at all; Diarrhoea/ vomiting grade 3= diarrhoea/ vomiting that prevented normal activity; Related= general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 46 | 33 | 33 | 112
Participants
  Any Diarrhoea/vomiting Dose 1 | 10 | 6 | 3 | 19
  Grade 3 Diarrhoea/vomiting Dose 1 | 1 | 1 | 0 | 2
  Related Diarrhoea/vomiting Dose 1 | 6 | 1 | 2 | 9
  Any Drowsiness Dose 1 | 10 | 9 | 5 | 24
  Grade 3 Drowsiness Dose 1 | 1 | 0 | 0 | 1
  Related Drowsiness Dose 1 | 8 | 7 | 5 | 20
  Any Irritability/fussiness Dose 1 | 21 | 14 | 9 | 44
  Grade 3 Irritability/fussiness Dose 1 | 3 | 0 | 0 | 3
  Related Irritability/fussiness Dose 1 | 19 | 10 | 8 | 37
  Any Loss of appetite Dose 1 | 9 | 12 | 6 | 27
  Grade 3 Loss of appetite Dose 1 | 0 | 1 | 0 | 1
  Related Loss of appetite Dose 1 | 5 | 8 | 5 | 18
  Any Fever (Axillary) Dose 1 | 4 | 6 | 4 | 14
  Grade 3 Fever (Axillary) Dose 1 | 0 | 2 | 0 | 2
  Related Fever (Axillary) Dose 1 | 3 | 5 | 3 | 11
  Any Diarrhoea/vomiting Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Any Diarrhoea/vomiting Dose 2 | 8 | 3 | 2 | 13
  Grade 3 Diarrhoea/vomiting Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Grade 3 Diarrhoea/vomiting Dose 2 | 0 | 0 | 0 | 0
  Related Diarrhoea/vomiting Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Related Diarrhoea/vomiting Dose 2 | 7 | 2 | 1 | 10
  Any Drowsiness Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Any Drowsiness Dose 2 | 8 | 12 | 7 | 27
  Grade 3 Drowsiness Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Grade 3 Drowsiness Dose 2 | 1 | 1 | 1 | 3
  Related Drowsiness Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Related Drowsiness Dose 2 | 8 | 10 | 7 | 25
  Any Irritability/fussiness Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Any Irritability/fussiness Dose 2 | 14 | 17 | 10 | 41
  Grade 3 Irritability/fussiness Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Grade 3 Irritability/fussiness Dose 2 | 1 | 3 | 0 | 4
  Related Irritability/fussiness Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Related Irritability/fussiness Dose 2 | 13 | 15 | 10 | 38
  Any Loss of appetite Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Any Loss of appetite Dose 2 | 8 | 6 | 9 | 23
  Grade 3 Loss of appetite Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Grade 3 Loss of appetite Dose 2 | 0 | 1 | 0 | 1
  Related Loss of appetite Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Related Loss of appetite Dose 2 | 8 | 5 | 8 | 21
  Any Fever (Axillary) Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Any Fever (Axillary) Dose 2 | 14 | 12 | 10 | 36
  Grade 3 Fever (Axillary) Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Grade 3 Fever (Axillary) Dose 2 | 2 | 3 | 1 | 6
  Related Fever (Axillary) Dose 2: number analyzed (Participants) | 45 | 33 | 33 | 111
  Related Fever (Axillary) Dose 2 | 14 | 12 | 10 | 36
  Any Diarrhoea/vomiting Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Any Diarrhoea/vomiting Dose 3 | 10 | 3 | 3 | 16
  Grade 3 Diarrhoea/vomiting Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Grade 3 Diarrhoea/vomiting Dose 3 | 1 | 0 | 0 | 1
  Related Diarrhoea/vomiting Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Related Diarrhoea/vomiting Dose 3 | 9 | 2 | 1 | 12
  Any Drowsiness Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Any Drowsiness Dose 3 | 16 | 6 | 10 | 32
  Grade 3 Drowsiness Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Grade 3 Drowsiness Dose 3 | 2 | 0 | 1 | 3
  Related Drowsiness Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Related Drowsiness Dose 3 | 16 | 6 | 7 | 29
  Any Irritability/fussiness Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Any Irritability/fussiness Dose 3 | 28 | 15 | 11 | 54
  Grade 3 Irritability/fussiness Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Grade 3 Irritability/fussiness Dose 3 | 7 | 0 | 2 | 9
  Related Irritability/fussiness Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Related Irritability/fussiness Dose 3 | 26 | 15 | 10 | 51
  Any Loss of appetite Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Any Loss of appetite Dose 3 | 16 | 12 | 9 | 37
  Grade 3 Loss of appetite Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Grade 3 Loss of appetite Dose 3 | 2 | 0 | 2 | 4
  Related Loss of appetite Dose 3: number analyzed (Participants) | 45 | 33 | 33 | 108
  Related Loss of appetite Dose 3 | 15 | 12 | 7 | 34
  Any Fever (Axillary) Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Any Fever (Axillary) Dose 3 | 20 | 15 | 19 | 54
  Grade 3 Fever (Axillary) Dose 3: number analyzed (Participants) | 45 | 30 | 33 | 108
  Grade 3 Fever (Axillary) Dose 3 | 3 | 5 | 3 | 11
  Related Fever (Axillary) Dose 3 | 19 | 15 | 18 | 52
  Any Diarrhoea/vomiting Across doses | 17 | 11 | 7 | 35
  Grade 3 Diarrhoea/vomiting Across doses | 1 | 1 | 0 | 2
  Related Diarrhoea/vomiting Across doses | 14 | 5 | 3 | 22
  Any Drowsiness Across doses | 22 | 18 | 12 | 52
  Grade 3 Drowsiness Across doses | 3 | 1 | 2 | 6
  Related Drowsiness Across doses | 21 | 17 | 12 | 50
  Any Irritability/fussiness Across doses | 35 | 23 | 15 | 73
  Grade 3 Irritability/fussiness Across doses | 10 | 3 | 2 | 15
  Related Irritability/fussiness Across doses | 35 | 23 | 14 | 72
  Any Loss of appetite Across doses | 22 | 18 | 14 | 54
  Grade 3 Loss of appetite Across doses | 2 | 2 | 2 | 6
  Related Loss of appetite Across doses | 19 | 17 | 14 | 50
  Any Fever (Axillary) Across doses | 29 | 19 | 21 | 69
  Grade 3 Fever (Axillary) Across doses | 5 | 8 | 4 | 17
  Related Fever (Axillary) Across doses | 28 | 19 | 20 | 67

25. Secondary Outcome: Number of Subjects With Medically-attended Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination. Analysis of intensity and relationship to vaccination of MAEs was not performed.
Time Frame: During the entire study period (from Day 0 to Day 364)
Population: The analysis was performed on the Total Vaccinated Cohort (TVC), which included all subjects with at least one vaccine administration documented. Analyses were done by age stratum and overall.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 46 | 34 | 33 | 113
Participants | 29 | 19 | 20 | 68

26. Secondary Outcome: Number of Subjects With Potential Immune-mediated Disease (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: During the entire study period (from day 0 to Day 364)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 46 | 34 | 33 | 113
Participants | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" was defined as an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination. "Grade 3" was defined as an AE which prevented normal, everyday activities. "Related" was defined as an AE assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 21 day follow-up period after each vaccination (Day 0 - Day 21, Day 21 - Day 42, Day 182 - Day 203)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 46 | 34 | 33 | 113
Participants
  Any AE(s) | 29 | 19 | 24 | 72
  Grade 3 AE(s) | 5 | 3 | 2 | 10
  Related AE(s) | 13 | 5 | 7 | 25

28. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: as for outcome 27
Time Frame: During an 84 day follow-up period after each vaccination (Day 0 - Day 84, Day 21 - Day 105, Day 182 - Day 266)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 46 | 34 | 33 | 113
Participants
  Any AE(s) | 32 | 23 | 22 | 77
  Grade 3 AE(s) | 4 | 4 | 2 | 10
  Related AE(s) | 9 | 3 | 6 | 18

29. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed included medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/ incapacity.
Time Frame: During the entire study period (from Day 0 to 364)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group | GSK1562902A Group
Number analyzed (Participants) | 46 | 34 | 33 | 113
Participants | 5 | 4 | 0 | 9

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 364; Solicited local and general symptoms: During the 7-day (Days 0-6) post-vaccination period; Unsolicited adverse events: During the 84-day (Days 0-84) post-vaccination period.
Groups:
- GSK1562902A 6 to 12 M Group: Subjects between 6 and 12 months of age, who received 2 primary doses of A/Indonesia/05/2005 GSK1562902A vaccine on Days 0 and 21 and 1 booster dose of the A/turkey/Turkey/1/2005 GSK1562902A vaccine on Day 182.
- GSK1562902A 12 to 24 M Group: Subjects between 12 and 24 months of age, who received 2 primary doses of A/Indonesia/05/2005 GSK1562902A vaccine on Days 0 and 21 and 1 booster dose of the A/turkey/Turkey/1/2005 GSK1562902A vaccine on Day 182.
- GSK1562902A 24 to 36 M Group: Subjects between 24 and 36 months of age, who received 2 primary doses of A/Indonesia/05/2005 GSK1562902A vaccine on Days 0 and 21 and 1 booster dose of the A/turkey/Turkey/1/2005 GSK1562902A vaccine on Day 182.
Arm/Group | GSK1562902A 6 to 12 M Group | GSK1562902A 12 to 24 M Group | GSK1562902A 24 to 36 M Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 5/46 | 4/34 | 0/33
Other Adverse Events (participants affected / at risk) | 45/46 | 32/34 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1562902A 6 to 12 M Group (N=46) | GSK1562902A 12 to 24 M Group (N=34) | GSK1562902A 24 to 36 M Group (N=33)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1562902A 6 to 12 M Group (N=46) | GSK1562902A 12 to 24 M Group (N=34) | GSK1562902A 24 to 36 M Group (N=33)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 8 (8) | 2 (6)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 22 (33) | 18 (30) | 14 (24)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 13 (16) | 6 (7) | 3 (5)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (2)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site scab (General disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 35 (63) | 23 (46) | 15 (30)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (8) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Pain (General disorders) | 27 (45) | 19 (33) | 21 (45)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 31 (45) | 20 (39) | 22 (40)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 5 (6) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 2 (2) | 3 (4)
Roseola (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 22 (34) | 18 (27) | 12 (22)
Swelling (General disorders) | 6 (8) | 6 (8) | 1 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 5 (7) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 5 (6) | 12 (14)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (30) | 11 (15) | 10 (12)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.